CLINICAL TRIAL: NCT05588076
Title: Predictive Factors of Endometrial Lesions in Patients With Abnormal Uterine Bleeding
Brief Title: Endometrial Lesions Predictions
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AUBEM
Record Dates: First submitted 2022-10-07; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Endometrial Neoplasms
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- normal endometrial
  Interventions: Other: no intervention
- endometrial lesions

INTERVENTIONS:
Other: no intervention — no intervention
  Groups: normal endometrial

SUMMARY:
To explore the risk factors of endometrial lesions in patients with abnormal uterine bleeding and establish prediction models which can discriminate between different endometrial etiologies of abnormal uterine bleeding(AUB).

ELIGIBILITY:
Inclusion Criteria:

* 1) non-pregnancy related abnormal uttering bleeding（AUB） in women of 18-60 years old; 2)women who had indications for hysteroscopy and endometrial histology in the study period

Exclusion Criteria:

* 1) postmenopausal women, 2) AUB due to other causes such as hormones or medications, coagulation disorders, and vascular malformation of the uterus; 3) final diagnosis outside the scope of this study.

Ages: 18 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: This cross-sectional study was approved by the Institutional Ethics Committee and conducted in the Beijing Friendship Hospital, Capital Medical University in China
Sampling Method: Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
pathology of endometrial lesions | 1 year
  Endometrial tissue was curettaged and sent for pathological examination in 10% formalin. A senior pathologist who was not blinded to clinical and ultrasound information examined the samples and determined the final diagnosis. The outcomes of histology are classified as normal endometrium and endometrial lesions, which include 1)endometrial polyps,2)endometrial hyperplasia without atypia, 3)endometrial atypical hyperplasia and 4) endometrial carcinoma.

SECONDARY OUTCOMES:
Ultrasonographic Examination | 1 year
  VS examinations were performed by an experienced physician with a vaginal probe of 5.5 MHz of a GE VolusonE10 Ultrasound device to look for endometrial thickness and abnormal echoes. Endometrial thickness (ET) was measured at the thickest part with double layers

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Zhang, Dr, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No